CLINICAL TRIAL: NCT00035490
Title: Efficacy and Safety Evaluation of Azimilide Dihydrochloride in Patients With Implantable Cardioverter Defibrillators
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Jose Brum, MD, Procter & Gamble Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000098
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — azimilide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo tablets
  Interventions: Drug: placebo
- 2 (Experimental): 75 mg azimilide
  Interventions: Drug: Azimilide Dihydrochloride
- 3 (Experimental): 125 mg azimilide
  Interventions: Drug: Azimilide Dihydrochloride

INTERVENTIONS:
Drug: Azimilide Dihydrochloride — 125 mg azimilide, once a day for one year
  Arms: 3
Drug: placebo — placebo tablet, once daily for one year
  Arms: 1
Drug: Azimilide Dihydrochloride — 75 mg azimilide, once a day for one year
  Arms: 2

SUMMARY:
Implantable cardioverter defibrillators (ICDs) have been developed to treat ventricular tachycardia or fibrillation (abnormal heart rhythms) by electrical shock or by pacing the heart. ICD therapy is established as highly effective for stopping life-threatening arrhythmias, but it does not preclude the use of anti-arrhythmic drugs for prevention and to decrease the frequency of ICD shocks.

The safety and effectiveness of oral azimilide dihydrochloride in reducing the frequency of ICD shocks has been investigated previously in a placebo-controlled study in patients with ICDs. These results need to be confirmed in this larger double-blind, placebo-controlled study with approximately 600 patients.

ELIGIBILITY:
Inclusion criteria:

* Currently have an ICD implanted
* Have had a documented episode of symptomatic arrhythmias that triggered a spontaneous ICD shock within 180 days of randomization.
* If the ICD implant is recent, the patient must have had a documented episode of sustained arrhythmias or cardiac arrest within 42 days before implantation of the ICD

Exclusion criteria:

* have severe heart failure
* have a current diagnosis of psychosis
* use illicit drugs
* abuse alcohol
* if female, are currently breast feeding, or plan to become pregnant during the study
* are currently taking antiarrhythmic drugs or other drugs that prolong the QTc interval (a measurement taken from the ECG)
* creatinine >2.5 mg/dL (221 mmol/L)
* potassium <4.0 mEq or >5.5 mEq
* have a neutrophil count (ANC) < 100 mL (low count of a type of white blood cell) at time of randomization
* have 2 or more consecutive QTc values >440 msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2001-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Reducing the recurrence of all-cause shocks plus symptomatic ATP | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Brum, MD, Study Director — Procter and Gamble
Locations (142):
- United States (78):
  - The Heart Group, Mobile, Alabama
  - Tri-City Cardiology Consultants, P.C., Mesa, Arizona
  - UAMS Dept of Cardiology, Little Rock, Arkansas
  - ATC/Cardio Medical Grp, Beverly Hills, California
  - Loma Linda Univ. Med. Ctr., Loma Linda, California
  - Good Samaritan Hospital, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Regional Cardiology Associates, Sacramento, California
  - Cardiac Arrythmia Associates, San Diego, California
  - UCSD Medical Center, San Diego, California
  - Memorial Hospital, Colorado Springs, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Arrythmia Consultants, Fort Lauderdale, Florida
  - Southwest Florida Health Group, Fort Myers, Florida
  - Jacksonville Heart Center, Jacksonville, Florida
  - The Watson Clinic, LLP, Lakeland, Florida
  - Univ. Miami Jackson Mem. med. Ctr., Miami, Florida
  - Florida Heart Institute, Orlando, Florida
  - Memorial Health Systems/Cardiology Research Associates, Ormond Beach, Florida
  - Loyola University Med. Ctr., Maywood, Illinois
  - University of Iowa Hospital, Iowa City, Iowa
  - Mid-America Cardiology c/o KU medical Ctr, Kansas City, Kansas
  - University Cardiology, Louisville, Kentucky
  - Louisville Cardiology Medical Group, PSC, Louisville, Kentucky
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Maine Cardiology Assoc., Portland, Maine
  - Mid-Atlantic Cardiovascular Associates, Baltimore, Maryland
  - St Elizabeth Medical Center, Boston, Massachusetts
  - Lahey Hitchcock Medical Ctr., Burlington, Massachusetts
  - Baystate Medical Center-Cardiology Research, Springfield, Massachusetts
  - University of Mass. Medical Ctr. Division of Cardiovascular Medicine, Worcester, Massachusetts
  - SMDC Education Research, Duluth, Minnesota
  - University of Minnesota-Cardiology, Minneapolis, Minnesota
  - Nevada Cardiology, Las Vegas, Nevada
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Atlantic Health Systems, Passaic, New Jersey
  - Arrhythmia and Pacemaker Consultants, West Orange, New Jersey
  - Brookdale University Hospital, Brooklyn, New York
  - Huntington Hospital, Huntington, New York
  - Cardiology Assoc., PC, Johnson City, New York
  - St. Lukes/Roosevelt Hospital Center, New York, New York
  - The Mt Sinai Medical Ctr., New York, New York
  - Rochester Cardiopulmonary Group, Rochester, New York
  - University of Rochester Strong mem. Hospital, Rochester, New York
  - Buffalo Cardiology & Pulmonary Assoc., Williamsville, New York
  - Mid Carolina Cardiology, Charlotte, North Carolina
  - Duke University Medical Ctr., Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - United HealthNetwork/Ohio Heart Center, Canton, Ohio
  - The Lindnar Clinical Trial Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Midwest Cardio Res. Foundation, Columbus, Ohio
  - Dayton Cardiac EP, Dayton, Ohio
  - Medical College of Ohio, Toledo, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Cardiovascular Assoc., Eugene, Oregon
  - Doylestown Medical Hospital, Doylestown, Pennsylvania
  - Hershey Med. Ctr.-Div. Cardiology, Hershey, Pennsylvania
  - Lancaster Heart Foundation, Lancaster, Pennsylvania
  - Univ of PA/Presbyterian Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Barry Alpert, MD, FACC, Pittsburgh, Pennsylvania
  - Blackstone Cardiology Assoc. P.C., Pawtucket, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - Mid-State Cardiology, Nashville, Tennessee
  - Heart Place/Baylor University of Medicine, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Medical Ctr., Salt Lake City, Utah
  - U. OF Virginia/Dept of Cardiology, Charlottesville, Virginia
  - The Cardiovascular Grp./Attn: Mandy Murphy, Fairfax, Virginia
  - Medical College of VA, Richmond, Virginia
  - Inland Cardiology/The Heart Inst., Spokane, Washington
  - Cardiology Associates of Green Bay, Green Bay, Wisconsin
  - Wisconsin Ctr for Clinical Research, Milwaukee, Wisconsin
- Belgium (2):
  - A.Z. Sint-Jan, Ruddershove, 10, Bruges
  - Clin. Univ. UCL de Mont-Godinne-, Yvoir
- Canada (11):
  - University of Alberta Hospital, Edmonton, Alberta
  - Cardiac Arrythmia Trials/Royal Jubilee Hosp., Victoria, British Columbia
  - Academisch ZiekenhuisRotterdam, Thoraxentrum Dr. Molewaterplein 40, Rotterdam, Newfoundland and Labrador
  - Health Sciences Ctr, St. John's, Newfoundland and Labrador
  - Isala Klinieken Loc Weezenlanden Afd. Cardiologie Groot Wezenland 20, Zwolle, Newfoundland and Labrador
  - QE II Health Sciences Ctr., Halifax, Nova Scotia
  - Hamilton General Hospital/McMaster Clinic, Hamilton, Ontario
  - St Michaels Hospital 30 Bond Street 7-050 Queen, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Laval Hospital, Ste-Foy, Quebec
  - Winnepeg Health Science Ctr., Winnepeg
- France (9):
  - CHRU de Lille-Hopital Cardiologique-Bd du Pr Leclerc, Lille
  - Centre hospitalier L. Pradel-28 av. du doyen Lepine, Lyon
  - Hopital Nord-Chemin Bourrely St Antoine, Marseille
  - CHRU de Nancy-29 av. de Lattre de Tassigny, Nancy
  - CHRU de Nantes-Hopital G. et R. Laennec-bd Jacques Monod, Nantes
  - Hopital Lariboisiere-2 rue A. Pare, Paris
  - Hopital cardiologique du Haut Leveque-av. de Magellan, Pessac
  - CHRU de Rennes-Hotel Dieu-2 rue l'hotel Dieu, Rennes
  - CHRU de TOURS-Hopital TROUSSEAU-Chanbray les Tours, Tours
- Germany (23):
  - Herz-kreislauf-Klinik Bevensen AG Kardiologie Akut Romstedter Str. 25, Bad Bevensen
  - Kerckhoff Klinik Abteilung Elektrophysiologie Benekestr. 2, Bad Nauheim
  - Herzzentrum NRW Kardiologische Ambulanz Georgstr. 11, Bad Oeynhausen
  - Krankenhaus Am Urban Innere Medizin I (Kardiologie) Dieffenbachstr. 1, Berlin
  - Charite Campus Buch Franz-Vollhard-Klinik Wiltbergstr. 50, Berlin
  - Virchow-Klinikum Franz-Volhard-Klinik Wiltbergstr. 50, Berlin
  - Universitatsklinikum Bonn Medizinische Klinik und Poliklinik II Sigmund-Freud-Str. 25, Bonn
  - Stadtisches Klinikum Brandenburg Medizinische Klinik I Kardiologie Hochstr. 29, Branderburg An Der Havel
  - Klinikum Coburg Ketschendorferstr. 33, Coburg
  - Evangelische Krankenhaus Abteilung Kardiologie Kirchfeldstr. 40, Düsseldorf
  - Universitatsklinikum Dusseldorf Klinik fur Kardiologie Moorenstr. 5, Düsseldorf
  - Klinikum der Johann-Wolfgang-Goethe-Universitat Medizinische Klinik IV Abteilung Elektrophysiologie Theodor-Stern-Kai 7, Frankfurt
  - Medizinische Universitatsklinik, Freiburg im Breisgau
  - Universitats-Krankenhaus Eppendorf Abteilung Kardiologie Martinistr. 52, Hamburg
  - Medizinische Universitats Klinik Heidelberg Medisin III (Kardiologie) Bergheimerstr. 58, Heidelberg
  - Klinikum der Stadt Ludwigshafen Bremserstr. 79, Ludwigshafen
  - Medizinische Universitatsklinik Leipzigerstr. 44, Magdeburg
  - Universitatsklinikum I. Medizinische Klinik Kardiologie/Angiologie/Pneumologie Theodor-Kutzer-Ufer 1-3, Mannheim
  - Deutsches Herzzentrum Minchen Lazarettstr. 36, München
  - Klinikum Grobhadern Universitat Munchen Marchioninistr. 15, München
  - Stadt. Klinikum Nurnberg-Sud Med. Klinik 8-Kardiologie Kardiologie KH II/8, Nuremberg
  - Medizinische Klinik und Poliklinik Universitat Tubingen Ottfried-Muller-Str. 10, Tübingen
  - Klinikum Wuppwrtal GmbH Klinik Fur Herz-und Thoraxchirugie Arrenbergerstr. 20, Wuppertal
- Italy (4):
  - Istituto di Malattie cardiovasolari policlinico di bari piazza G Cesare 11, Bari
  - Ospedale Maggiore della carita II Divisione di cardiologia, corso mazzini 18, Novara
  - Policlinico Matteo Dippartimento di cardiologia Pizza Golgi, 2, Pavia
  - Divisione di cardiologia Ospedale s. Flippo Neri, Via Martinotti 20, Roma
- Netherlands (5):
  - Academisch Medisch Centrum Amsterdam Afd. Cardiologie Meibergdreef 9, Amsterdam
  - Catharina Ziekenhuis Afd. Cardiologie Postbus 1350, Eldhoven
  - Academisch Ziekenhuis Groningen Thoraxcentrum Hanzeplein 1, Groningen
  - Leids Universitair Medisch Centrum Afd. Cardiologie Postbus 9600, Leiden
  - SintAntonius Ziekenhuis Afd R&D Cardiologie Koekoekslaan 1, Nieuwegein
- Poland (5):
  - ll Klinika Chorob Serca Akademii Medycznej w Gdansku Kieturakisa 1, Gdansk
  - 1 Klinka kardiologii Slaska Akademia Medyczna, Ziolowa 47, Katowice
  - Oddzial kardiologii-Instut kardiologii, Ul Powstancow, Szczecin
  - Instytut Kardiologii Klinika Choroby Wiencowej,ul Spartanka 1, Warsaw
  - Instytut Kardiologii-Klinka Kardiologii Ogolnej, ul. Alpejska 42, Warsaw
- Spain (5):
  - Hospital Clinic i Provincial, Servicio de Cardiologia, Villarroel, 170, Barcelona
  - Clinica Puerta de Hierro, San Martin de Porres, 4, Madrid
  - Hospital 12 de Octubre, Carretera de Andalucia, km. 5, 4, Madrid
  - Hospital Virgen de la Victoria, Campus Universitario de Teatinos, s/n, Málaga
  - Hospital Clinico Universitario de Valencia, Avenida Blasco Ibanez, 17, Valencia